CLINICAL TRIAL: NCT01212861
Title: Surgical Treatment of Refractory Open Angle Glaucoma - A Prospective, Open-Label, Pilot Study
Brief Title: Surgical Treatment of Refractory Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iScience Interventional Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060410
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suprachoroidal Dissection Instrument (Experimental)
  Interventions: Device: Suprachoroidal Dissection Instrument (SDI)

INTERVENTIONS:
Device: Suprachoroidal Dissection Instrument (SDI) — The Suprachoroidal Dissection Instrument (SDI) is a manually operated, non-powered, re-usable ophthalmic surgical instrument. The SDI is designed to enter a surgically exposed Schlemm's canal and be advanced up to 90 degrees around the canal from the entry site.
  Other Names: SDI

SUMMARY:
The primary objective of this study is to evaluate the safety, efficacy, and performance of the Suprachoroidal Dissection Instrument in creating a fistula between Schlemm's canal and the suprachoroidal space in refractory, open angle glaucoma subjects.

DETAILED DESCRIPTION:
The Suprachoroidal Dissection Instrument (SDI) is a manually operated surgical instrument designed for use within Schlemm's canal. The instrument can access Schlemm's canal through a small ab-externo dissection, allowing use in eyes with scarring due to previous surgery or trauma.

ELIGIBILITY:
Inclusion Criteria:

* Available for up to 3 years follow-up.
* Diagnosed with primary open-angle, pseudoexfoliative, or pigmentary glaucoma or more than one glaucoma diagnosis of these types.
* Subject scheduled to undergo glaucoma surgery with the Suprachoroidal Dissection Instrument involving creation of fistula between Schlemm's canal and the suprachoroidal space without combined cataract surgery.
* Subject has failed at least one incisional glaucoma surgery (trabeculectomy, tube shunt, deep sclerectomy, viscocanalostomy, canaloplasty) or angle surgery (Trabectome) OR Is not a candidate for conventional glaucoma surgery due to reasons such as the presence of scleral buckle or compromised conjunctiva.
* Subject has IOP ≥ 16 mm Hg on maximally tolerated medications within the six week (-42 days) period prior to surgery.
* Visual field defect defined as mean deviation (MD) score worse than or equal to -10 dB on the Swedish Interactive Threshold Algorithm [SITA] Standard 24-2 Humphrey Analysis during the 6 month period prior to surgery. OR Subject has vertical cup-to-disk ratio ≥ 0.75 during the 6 month period prior to surgery.

Exclusion Criteria:

* Significant lens opacities or patient is candidate for cataract surgery during the duration of the study.
* The patient had developmental glaucoma or a secondary glaucoma including steroid-induced, uveitic, or neovascular glaucoma (with the exception of pigmentary and pseudoexfoliative glaucoma).
* The patient has narrow angle component possibly associated with glaucoma in the operative eye.
* The subject has angle recession in the operative eye.
* Significant ocular disease other than glaucoma affecting the assessment of visual function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Postoperative intraocular pressure, glaucoma medication usage, and visual acuity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Fellman, MD, Principal Investigator — Glaucoma Associates of Texas
Locations (1):
- Glaucoma Associates of Texas, Dallas, Texas, United States